CLINICAL TRIAL: NCT02200627
Title: Forxiga Tablets Specific Clinical Experience Investigation for Elderly
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1692C00015
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Diabetes; Forxiga; Elderly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the investigation is to confirm the following under the post-marketing actual use of Forxiga Tablets (hereinafter referred to as Forxiga) in elderly patients.

* Development of ADRs specified as Key Investigation Items and the risk factors
* Contributing factors possibly having an impact on the safety and efficacy
* Development of ADRs unexpected from the Precautions for use and ADRs under actual drug use

ELIGIBILITY:
Inclusion Criteria:

Patients treated with Forxiga for the first time during three months after the launch due to type 2 diabetes mellitus, which is the indication of the drug, aged 65 or over at the time when Forxiga was started.

In addition, patients receiving the study drug of Forxiga before the launch should be included also.

Exclusion Criteria: N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with Forxiga for the first time during three months after the launch due to type 2 diabetes mellitus, which is the indication of the drug, aged 65 or over at the time when Forxiga was started.
  In addition, patients receiving the study drug of Forxiga before the launch should be included also.
Sampling Method: Non-Probability Sample
Enrollment: 1724 (Actual)
Dates: Start 2014-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Adverse event incidence | from baseline to 1 year

CONTACTS AND LOCATIONS:
Locations (46):
- Japan (46):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagawa
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Miyazaki
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Niigata
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokushima
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Toyama
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yamaguchi
  - Research Site, Yamanashi

REFERENCES:
- See also: CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2993&filename=Synopsis_D1692C00015.pdf